CLINICAL TRIAL: NCT01360593
Title: Induction Gemcitabine/Capecitabine Followed by SBRT in Pancreatic Adenocarcinoma A Prospective Evaluation in Patients With Locally Advanced Pancreas Cancer
Brief Title: Gemcitabine/Capecitabine Followed by SBRT in Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David A. Clump, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, David A. Clump, MD, PhD, Assistant Professor, Radiation Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-139
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Capecitabine; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Gem, Xeloda, SBRT (Other)
  Interventions: Drug: Gemcitabine; Drug: Capecitabine; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be administered for 2 weekly doses every 3 weeks commencing 12 weeks prior to stereotactic radiosurgery as follows:
  Gemcitabine 1,000 mg/m2 IV over 30 minutes on Day 1, and 8 of 21- day cycle. This will be done for up to 4 cycles.
  Other Names: Gemzar
Drug: Capecitabine — Capecitabine will be taken orally twice daily on days 1-14 every 3 weeks for 4 cycles (12 weeks) prior to stereotactic radiosurgery as follows:
  Capecitabine 650 mg/m2 twice daily for days 1-14 every 3 weeks for up to 4 cycles.
  Other Names: Xeloda
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Fractionated SBRT will be delivered to patients that have stable disease, partial response, or complete response after chemo in the following manner:
  12 Gy x 3 fractions (36 Gy total) This will be given every other day.
  Other Names: CyberKnife; Trilogy; True Beam; Radiosurgery; SBRT

SUMMARY:
The current study seeks to further investigate the impact of up-front systemic therapy in combination with fractionated SBRT for potentially resectable, locally-advanced pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
All subjects will have a baseline CT or FDG-PET/CT prior to initiation of therapy. This will be done at the Hillman or in Radiation Oncology. Enrolled patients will undergo appropriate lab work and staging as described

1. Albumin, alkaline phosphatase, glucose, electrolytes
2. Ca 19-9 and CEA
3. Due to an interaction of capecitabine and oral coumadin-derivative anticoagulants and risk of bleeding/thrombotic events, if a patient is on coumadin, frequent monitoring of INR and dose adjustments of anticoagulants must be exercised during protocol treatment. Alternatively, low molecular weight heparin may be substituted for oral anticoagulants Chemotherapy will be initiated consisting of gemcitabine 1000mg/m2 IV on day 1 and 8 of a 21 day cycle. Dosage for gemcitabine is described below using the Body surface area (BSA).

BSA will be calculated from body weight in kg, recorded prior to every gemcitabine dosing, and height in cm, recorded at baseline.

Premedication for Gemcitabine

A standard, FDA-approved antiemetic medication will be administered to study participants at the discretion of the treating oncologist (investigator) one-half hour prior to the gemcitabine infusion. Examples of standard antiemetics include ondansetron (Zofran), granisetron (Kytril), dolasetron (Anzemet), compazine, and dexamethasone. The dosage and route of administration will be determined by the treating oncologist based upon the given clinical scenario.

In addition, capecitabine 650mg/m2 PO will be taken twice daily on days 1-14 of a 3 week cycle. Four cycles total (12 weeks) of chemotherapy will be given. Dosage for capecitabine is described below using the Body surface area (BSA).

BSA will be calculated from body weight in kg, recorded prior to every capecitabine dosing, and height in cm, recorded at baseline.

Capecitabine (Xeloda; F. Hoffmann-La Roche AG, Basel, Switzerland) is supplied as ﬁlm-coated tablets in two dose strengths (150 and 500 mg); the closest practical dose (by rounding up or down) calculated on body-surface area based on a combination of tablets is taken within 30 minutes after the end of a meal.

Patients will be assessed during chemotherapy with appropriate dose modifications made based on toxicity. Following the completion of chemotherapy, a new FDG-PET/CT or CT will be obtained to assess response and plan for SBRT. For those patients with SD, PR, or CR, SBRT will be planned and delivered.

Fidiucial placement In addition, all patients will have fiducial markers placed for localization at time of SBRT. Three to five soft-tissue fiducials (markers) will be placed in and/or around the tumor, at least 1cm apart. Oftentimes, these are placed at the time of endoscopic ultrasound and biopsy for diagnosis. If that is not the case, patients will be scheduled for a repeat EUS and have the markers placed prior to CT or FDG-PET/CT simulation. Alternatively, fiducials may be placed at the time of staging laparoscopy.

Stereotactic Body Radiotherapy Planning SBRT will be done in Shadyside Radiation Oncology.

An SBRT plan will be created based on the disease contoured on the CT and PET. The plan will be to deliver fractionated SBRT to the isodose line best encompassing the PTV:

12 Gy x 3 fractions (36 Gy total)

Careful evaluation of the each plan will be conducted by the radiosurgical team to ensure that normal tissues and critical structures tolerances are maintained.

The maximum dose (in Gy) within the treatment volume (MD), prescriptions dose (PD), and the ratio of MD/PD (as a measure of heterogeneity within the target volume), prescription isodose volume (PIV in mm3), tumor volume (TV in mm3), and the ratio of PIV/TV (as a measure of dose conformity of the treatment relative to the target) will be recorded.

Quality of Life Assessment Quality of life assessment using the Functional Assessment of Cancer Therapy - General (FACT-G) tool, which is a validated tool, will be administered to all subjects prior to treatment and at each follow-up visit.

For patients with potentially resectable tumors, they will be assessed 10 - 12 weeks after SBRT by a multidisciplinary team including two expert pancreas surgeons and by FDG-PET/CT or CT scan. If deemed appropriate, patients with an adequate response will be taken for surgical resection. This will be performed as standard care.

Time frames for chemotherapy and SBRT for 4 cycles of gemcitabine and capecitabine. The SBRT will not start until twelve weeks after the chemotherapy stops and will last approximately one week. Each cycle of gemcitabine and capecitabine is three weeks. Upon completion of treatment patients will be followed for survival for 24 months. They will be in the study for approximately two years give or take a few months.

Interim medical history and physical examination 4 - 6 weeks after SBRT.

Serum chemistry and electrolytes to include BUN, creatinine, sodium, potassium, bicarbonate, chloride, calcium, magnesium, glucose, total bilirubin, AST, ALT, alkaline phosphatase prior to chemotherapy treatments, 4 -6 weeks post-SBRT treatment, and then at follow-up as clinically indicated

Hematologic studies to include CBC with differential and platelet count weekly during chemotherapy sessions and then repeated 4-6 weeks post-SBRT treatment and then at follow-up as clinically indicated

CT or FDG-PET/CT scans (for consistency procedure done at screening/planning will continue in follow-up) will be obtained at 10-12 weeks post-treatment and will be reviewed for evidence of response. Subjects who demonstrate no evidence of distant metastases and meet RECIST criteria of partial response, complete response, or stable disease will be offered surgical exploration and attempted curative resection. Subjects demonstrating unresectable disease or progression of disease will be started on systemic chemotherapy at the discretion of the treating medical oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the pancreas
* Subjects will be staged according to the 2010 AJCC staging system with pathologic stage T1-4, N0-1 being eligible; and have a primary tumor of the pancreas (i.e., pancreatic head, neck, uncinate process, body/tail
* Tumor must be deemed to be borderline resectable or locally advanced by radiographic criteria defined by Varadhachary et al.26 Final CT confirmation of surgical staging/eligibility will be by two expert pancreatic surgeons
* Disease confined to locoregional site confirmed by FDG-PET/CT or CT and diagnostic staging laparoscopy to ensure no occult peritoneal implants
* Disease must be encompassed in a reasonable SBRT "portal" as defined by the treating radiation oncologist
* Measurable disease on imaging studies (MRI, CT, FDG-PET/CT or physical exam), including maximum diameter/dimension, must be present for assessment of response
* Karnofsky performance status > 70 (ECOG 0-1)
* Age > 18
* Estimated life expectancy > 12 weeks
* Patient must have adequate renal function as defined by serum creatinine<1.5mg/dl obtained within 28 days prior to registration
* Patient must have adequate bone marrow function as defined by absolute neutrophil count>1500/mcl and platelets>100,000/mcl, obtained within 28 days prior to registration
* Patient must have adequate hepatic function as defined by total bilirubin <1.5 x IULN(institutional upper limit of normal) and either SGOT or SGPT <2.5x IULN, obtained within 28 days prior to registration.
* Patient must be able to swallow enteral medications. Patient must not require a feeding tube. Patient must not have intractable nausea or vomiting, GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, or uncontrolled inflammatory bowel disease (Chron's, ulcerative colitis).
* Diabetes must be controlled prior to FDG-PET/CT scanning (blood glucose <200 mg/dL)
* Ability to provide written informed consent
* Patient must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, history of myocardial infarction or cerebrovascular accident within 3 months prior to registration, uncontrolled diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not be pregnant because of the risk of harm to the fetus. Nursing women may participate only if nursing is discontinued, due to the possibility of harm to nursing infants from the treatment regimen. Women/men of reproductive potential must agree to use an effective contraception method.

Exclusion Criteria:

* Non-adenocarcinomas, adenosquamous carcinomas, islet cell carcinomas, cystadenomas, cystadenocarcinomas, carcinoid tumors, duodenal carcinomas, distal bile duct, and ampullary carcinomas are not eligible.
* Evidence of distant metastasis on upright chest x-ray (CXR), computed tomography (CT) or other staging studies
* Subjects with recurrent disease
* Prior radiation therapy to the upper abdomen or liver
* Prior chemotherapy
* Subjects in their reproductive age group should use an effective method of birth control. Subjects who are breast-feeding, or have a positive pregnancy test will be excluded from the study
* Any co-morbidity or condition of sufficient severity to limit full compliance with the protocol per assessment by the investigator
* Concurrent serious infection
* Previous or current malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in situ, adequately treated basal cell or squamous cell carcinoma of the skin, and treated low-risk prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-07-25 (Actual); Primary Completion 2016-03-13 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Clump, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Gem + Xeloda + SBRT: Gemcitabine administered for 2 weekly doses every 3 weeks commencing 12 weeks prior to stereotactic radiosurgery as follows:
  Gemcitabine 1,000 mg/m2 IV over 30 minutes on Day 1, and 8 of 21- day cycle. This will be done for up to 4 cycles.
  Capecitabine taken orally twice daily on days 1-14 every 3 weeks for 4 cycles (12 weeks) prior to stereotactic radiosurgery as follows:
  Capecitabine 650 mg/m2 twice daily for days 1-14 every 3 weeks for up to 4 cycles.
  Fractionated Stereotactic Body Radiation Therapy (SBRT) delivered to patients that have stable disease, partial response, or complete response after chemo as 12 Gy x 3 fractions (36 Gy total) - Given every other day.
Period: Overall Study
Arm/Group | Gem + Xeloda + SBRT
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients that received study treatment.
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.49 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status [Count of Participants; unit: Participants] — he ECOG Performance Status is a measure of functional status, with scores ranging from 0-4. Scores: 0 = Fully active; no performance restrictions; 1 = Strenuous physical activity restricted; fully ambulatory and able to carry out light work; 2 = Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours; 3 = Capable of only limited self-care; confined to bed or chair >50% of waking hours; 4 = Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    ECOG Score of 0 | 14
    ECOG Score of 1 | 20
Karnofsky Performance Status [Mean (Standard Deviation); unit: units on a scale] — The Karnofsky Performance Status (KPS) scores range 0 - 100. Higher KPS scores means the patient is better able to carry out daily activities, used to determine a patient's prognosis, and used to measure changes in a patient's overall ability to function.
  units on a scale | 89.12 (9.65)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.10 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Local Progression-free Survival (LPFS)
Description: LPFS is defined as the time from enrollment to first documentation of progressive disease (PD) in the target lesion. For patients that undergo surgical resection, local progression will be defined as disease recurrence detected on follow-up imaging (CT or FDG-PET/CT) that is located within the SBRT target volume. Death or development of distant disease is not regarded as an event. Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.0, progressive disease is defined as at least a 25% increase in the longest diameter of a lesion, taking as reference the longest diameter recorded since the treatment started.
Time Frame: Up to 32 months
Population: Patients able to be evaluated for response after study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 34
months | 22.30801 [17.31417 to NA] — Upper bound of 95% CI not reached due to insufficient number of participants with events.

2. Secondary Outcome: Objective Response Rate (ORR) (Neoadjuvant Chemotherapy)
Description: Percentage of participants with response per RECIST v1.0. Per RECIST v1.0: Complete Response (CR): the disappearance of a lesion; Near Complete Response (NCR): at least an 80% decrease in the longest diameter of a lesion, taking as reference the longest diameter recorded since the treatment started. Partial Response (PR): at least a 30% decrease in the longest diameter of a lesion, taking as reference the longest diameter recorded since the treatment started.
Time Frame: Up to 24 months
Population: Patients receiving neoadjuvant chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 31
percentage of participants | 28.13

3. Secondary Outcome: Objective Response Rate (ORR) (Surgery After Chemotherapy and SBRT)
Description: as for outcome 2
Time Frame: Up to 24 months
Population: Patients treated with surgery after chemotherapy and SBRT.
Measure: Number; unit: percentage of participants
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 10
percentage of participants | 20.0

4. Secondary Outcome: Overall Survival (OS)
Description: The (median) length of time from enrollment to confirmed death from any cause.
Time Frame: Up to 32 months
Population: Patients that received study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 34
months | 18.82546 [13.86448 to NA] — Upper bound of 95% CI not reached due to insufficient number of participants with events.

5. Secondary Outcome: Time to Progression (TTP)
Description: The (median) length of time from enrollment to disease progression per Response Evaluation Criteria in Solid Tumors (v1.0). Per RECIST, Progressive Disease (PD) is defined at least a 25% increase in the longest diameter of a lesion, taking as reference the longest diameter recorded since the treatment started. For lesions without size response the maintenance of CA 19-9 level above the normal limits indicates disease progression.
Time Frame: Up to 5 years
Population: Patients that received study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 34
months | 16 [8.375 to 23.625]

6. Secondary Outcome: The Functional Assessment of Cancer Therapy - General (FACT-G)
Description: The Functional Assessment of Cancer Therapy - General (FACT-G) is a self-administered, 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. Quality of Life (QOL) evaluation will be administered prior to SBRT, after completion of SBRT, and at each follow-up. Scaling of items: Five-point scale for each questions from 0 (not at all) to 4 (very much); overall scoring 0-108. Higher scores indicated better quality of life.
Time Frame: Baseline; 2 - 4 weeks post chemotherapy; 4-6 weeks post SBRT; after surgery (up to 24 months)
Population: Treated patients that completed FACT/Quality of Life surveys.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 34
score on a scale
  Baseline | 54.0 [52.00 to 57.0]
  2-4 weeks after Chemo | 54.0 [0 to 62]
  4-6 weeks after SBRT | 51.5 [0 to 67]
  after Surgery, up to 24 months | 49.5 [0 to 61]

7. Secondary Outcome: Number of Participants Able to Undergo a Margin-negative Resection After Neoadjuvant Therapy
Description: Number of patients that are able to undergo a margin-negative resection after neoadjuvant therapy. Surgical evaluation: pathology records reviewed by operating surgeon to determine margin status as negative (not close (1-2.5mm), microscopically positive, and/or grossly positive).
Time Frame: Up to 24 months
Population: Patients that received study treatment with resection after neoadjuvant therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 35
Participants | 11

8. Secondary Outcome: Acute Toxicities Associated With SBRT
Description: Percentage of patients that experience treatment-related toxicities as graded according to Common Terminology Criteria for Adverse Events (CTCAE v4), within 3 months after treatment, by grade. Patients were monitored for potential toxicity throughout treatment.
Time Frame: Up to 3 months following SBRT treatment
Population: Patients that received SBRT.
Measure: Number; unit: percentage of participants
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 34
percentage of participants
  Grade 1 | 88.24
  Grade 2 | 29.41
  Grade 3 | 14.71
  Grade 4 | 2.94

9. Secondary Outcome: Late Toxicities Associated With SBRT
Description: Percentage of patients that experience treatment-related toxicities as graded according to Common Terminology Criteria for Adverse Events (CTCAE v4), greater than 3 months after treatment, by grade. Patients were monitored for potential toxicity throughout treatment.
Time Frame: From 3 months following SBRT treatment up to 24 months
Population: Patients that received study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 35
percentage of participants | 0

10. Secondary Outcome: Role of FDG-PET/CT
Description: 18F-FDG response measured using European Organization for Research and Treatment of Cancer (EORTC) 1999. Number of patients with non-FDG avid tumors with response to therapy using semi-quantitative SUV (standard uptake value) analysis based on lean body mass and/or body surface area is used in determining 18F-FDG uptake. [18F]-FDG uptake may provide an early, indication of the tumoricidal effect of anticancer agents.
Time Frame: Up to 24 months
Population: Due to a lack of insurance coverage for PET-CT in the context of pancreatic cancer, most insurers denied PET- CT in these patients, as such and to prevent any undue burden on patients, FDG-PET scans were not performed
Arm/Group | Gem + Xeloda + SBRT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 32 months for the study population.
Description: Adverse Events and Serious Adverse Events determined using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 Adverse Events were Grade 1 and Grade2 toxicities; Serious Adverse Events were Grade 3 and Grade 4 toxicities.
Arm/Group | Gem + Xeloda + SBRT
All-Cause Mortality (participants affected / at risk) | 30/34
Serious Adverse Events (participants affected / at risk) | 6/34
Other Adverse Events (participants affected / at risk) | 28/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gem + Xeloda + SBRT (N=34)
Neutropenia (Blood and lymphatic system disorders) | 2
White blood cell decreased ( leukopenia) (Investigations) | 2
Abdominal Infection (Infections and infestations) | 1
Ileus (Gastrointestinal disorders) | 1
Bleeding (Injury, poisoning and procedural complications) | 1
Stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gem + Xeloda + SBRT (N=34)
Neutropenia (Blood and lymphatic system disorders) | 6
Anemia (Blood and lymphatic system disorders) | 7
Liver Dysfunction (Hepatobiliary disorders) | 4
Hand-Foot (Infections and infestations) | 3
White blood cell decreased ( leukopenia) (Investigations) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Diarrhea (Gastrointestinal disorders) | 5
Edema (General disorders) | 1
Dermatitis (Injury, poisoning and procedural complications) | 1
Mucositis (General disorders) | 1
Platelet count decreased ( Thrombocytopenia) (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes